CLINICAL TRIAL: NCT01723618
Title: An Open-label, Randomised, Uncontrolled Trial Investigating the Pharmacokinetics of CRD007 After Single Dose Administration to Subjects With Abdominal Aortic Aneurysm (AAA)
Brief Title: Pharmacokinetics of CRD007 in Patients With Abdominal Aorta Aneurisms.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RSPR Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Cardoz-005
Record Dates: First submitted 2012-11-01; First posted 2012-11-08 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Abdominal Aortic Aneurisms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRD007 10 mg (Experimental): CRD007, 10 mg tablet, single dose
  Interventions: Drug: CRD007
- CRD007 25 mg (Experimental): CRD007, 25 mg tablet, single dose
  Interventions: Drug: CRD007
- CRD007 40 mg (Experimental): CRD007, 40 mg tablet, single dose
  Interventions: Drug: CRD007

INTERVENTIONS:
Drug: CRD007

SUMMARY:
The purpose of the study is to determine the plasma levels of CRD007 in patients with abdominal aortic aneurysms after the administration of single doses of tablets containing 10, 25 and 40 mg CRD007.

ELIGIBILITY:
Inclusion Criteria:

* Infra-renal abdominal aortic aneurysm

Exclusion Criteria:

* Significant concurrent disease or medical conditions that are deemed to interfere with the pharmacokinetics or the safety of CRD007 conduct of the trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - maximum plasma concentration (Cmax) | Pre-dose and until 12 hours post-dose
  Plasma concentrations of CRD007 will be measured and standard pharmacokinetic parameters as Cmax will be measured
Pharmacokinetics - time to maximum plasma concentration (tmax) | Pre-dose til 12 hours post-dose
  Plasma concentrations of CRD007 will be measured and standard pharmacokinetic parameters as tmax will be measured.
Pharmacokinetics - Area under the plasma concentration curve (AUC) | Pre-dose until 12 hours post-dose
  Plasma concentrations of CRD007 will be measured and standard pharmacokinetic parameters as AUC will be measured.
Pharmacokinetics - elimination half life (t1/2) | pre-dose until 12 hours post-dose
  Plasma concentrations of CRD007 will be measured and standard pharmacokinetic parameters as t1/2 will be measured

SECONDARY OUTCOMES:
Dose linearity | Pre-dose and until 12 hours post-dose
  Evaluation of dose linearity in the dose range 10 - 40 mg
Potential for accumulation | Pre-dose untill 12 hours post-dose
  To estimate the accumulation of CRD007 in the dose range 10 - 40 mg

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj F Groendal, MD, Principal Investigator — Department of Vascular Surgery Viborg Hospital Heiberg Allé 4 DK-8800 Viborg Denmark
Locations (1):
- Department of Vascular Surgery Viborg Hospital, Viborg, Denmark, Denmark